CLINICAL TRIAL: NCT06974474
Title: Potential Role of Guselkumab in Modulating PAIN Perception and Related Gene Pathways: a Proof-of-concept Study
Acronym: GUPAIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNTO1959PSA4016
Record Dates: First submitted 2024-09-25; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis Arthritis
Keywords: Guselkumab
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Psoriatic Arthritis (Other): Patients with Psoriatic Arthritis undergoing Guselkumab treatment
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab

SUMMARY:
Psoriatic arthritis (PsA) is a chronic musculoskeletal disease that affects 0.1%-1% of the general population and about 20% of patients with psoriasis. Patients with PsA have a multifaceted pain experience, which depends on various factors, including joint inflammation, as well as peripheral and central pain sensitization. Although chronic pain is the most common symptom of PsA, few is known about the mechanisms driving it. From this point of view, the interactions between immune cells and nociceptors in the context of inflammation-related pain are emerging as a hot topic. Many studies suggested that IL-23/IL-17 pathway may play a pivotal role in this regard. This is consistent with data currently available regarding Guselkumab in PsA. Indeed, according to DISCOVER 1 and DISCOVER 2, two randomized phase III trials, patients receiving Guselkumab achieved, among others, minimal disease activity state, significant improvement in the SF-36 physical component score, and visual analog scale of pain. This study proposal aims to evaluate the potential role of Guselkumab in modulating pain perception in PsA patients from a molecular, cellular, and electrophysiological point of view.

ELIGIBILITY:
Inclusion Criteria:

* A man or a woman at least 18 and no more than 80 years of age;
* Have a diagnosis of psoriatic arthritis (PsA) for at least 6 months the enrolment and meet Classification criteria for Psoriatic Arthritis (CASPAR) at screening;
* Inadequate response or intolerance of standard treatment (namely, methotrexate and/or TNF inhibitors);
* At least 3 months of non-biologic DMARDs (limited to methotrexate ≤25 mg/week, sulfasalazine ≤3 g/day, hydroxychloroquine ≤400 mg/day, and leflunomide ≤20mg/day) or at least 4 weeks of NSDAIDs for psoriatic arthritis;
* Patient eligible for Guselkumab (both monotherapy or combination therapy with methotrexate) treatment according to international recommendations, national and regional regulatory authorities, and EMA datasheet;
* VAS pain major than 15 mm at the enrolment;
* DAPSA major than 14 at the enrolment;
* Have at least 1 of the PsA subsets: oligoarticular or polyarticular PsA subset, distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, spondylitis with peripheral arthritis;
* Peripheral tender joints ≥ 1
* Peripheral swollen joints ≥ 1
* C-reactive protein ≥ 0.3 mg/dL
* Involvement (namely, swollen joint) of wrists or knees;
* Subjects naïve to bDMARDs or previously treated with up to 2 anti-tumor necrosis factor (TNFα) agents, discontinued for lack of benefit to an anti-TNFα therapy, as assessed by the treating physician, after at least 12 weeks of etanercept, adalimumab, golimumab, or certolizumab pegol therapy (or biosimilar) and/or at least a 14-week dosage regimen (i.e., at least 4 doses) of infliximab (or biosimilar). Documented lack of benefit may include inadequate improvement in joint counts, physical function, or disease activity; Intolerance to an anti-TNFα biologic therapy, as assessed by the treating physician, to etanercept, adalimumab, golimumab, certolizumab pegol, or infliximab (or biosimilars); If no intolerance or lack of benefit, the reason for discontinuation must be documented;
* If currently using non-biologic DMARDs (limited to methotrexate [MTX], sulfasalazine [SSZ], hydroxychloroquine [HCQ], or leflunomide [LEF]), subjects should have started treatment at least 3 months and the dose must be stable for at least 4 weeks before the first administration of study agent and should have no serious toxic side effects attributable to the non-biologic DMARD. If currently not using a MTX, SSZ, or HCQ, must have not received for at least 4 weeks before the first administration of study agent. If currently not using LEF, must not have received for at least 12 weeks before the first administration of study agent. If using MTX, the route of administration and dose must be stable and the dose must be ≤25 mg/week. If receiving SSZ, the dose must be ≤ 3g/day. If receiving HCQ, the dose must be ≤400 mg/day. If receiving LEF, the dose must be ≤20 mg/day.
* If currently using NSAIDs or other analgesics for PsA, subjects must be on a stable dose for at least 2 weeks before the first administration of study agent. If currently not using NSAIDs or other analgesics for PsA, must not have received NSAIDs or other analgesics for PsA within 2 weeks before the first administration of study agent;
* Are willing to refrain from the use of complementary therapies for PsA or psoriasis including ayurvedic medicine, traditional Taiwanese, Korean, or Chinese medications, and acupuncture within 2 weeks before the first study agent administration and through Week 52;
* Signed informed consent.

Exclusion Criteria:

* Diagnosis of fibromyalgia according to ACR 2016 criteria;
* Subjects with inflammatory diseases that might confound the evaluations of benefit of Guselkumab therapy, including but not limited to RA, axial spondyloarthritis (this does not include a primary diagnosis of PsA with spondylitis), systemic lupus erythematosus, or Lyme disease;
* Patients who received more than 2 anti-TNFα agents; - Has received an anti-TNF agent within the following timeframes: Infliximab (or its biosimilars) or golimumab (intravenous) within 8 weeks before the first administration Guselkumab; Golimumab (subcutaneous), adalimumab (or its biosimilars) or certolizumab pegol within 6 weeks before the first administration of study agent; Etanercept (or its biosimilars) within 4 weeks before the first administration of study agent;
* Has previously been treated with Guselkumab; - Diagnosis of psychiatric disorder according to DSM-V; - Pregnancy or lactation;
* Systemic or intra-articular glucocorticoids in the last 3 months;
* Has previously received any biologic treatment (other than anti-TNFα agents), including, but not limited to ustekinumab, abatacept, secukinumab, tildrakizumab, ixekizumab, brodalumab, risankizumab, or other investigative biologic treatment;
* Has previously received tofacitinib, baricitinib, filgotinib, peficitinib (ASP015K), decernotinib (VX-509), or any other Janus kinase (JAK) inhibitor, as well as apremilast;
* Has previously received any systemic immunosuppressants (e.g., azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus) within 4 weeks of the first administration of study agent;
* Has received non-biologic DMARDs (other than MTX, SSZ, HCQ, LEF) including, but not limited to chloroquine, gold preparations, and penicillamine within 4 weeks before the first administration of study agent;
* Is currently receiving 2 or more allowed non-biologic DMARDs at baseline;
* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic (with the exception of PsA), genitourinary, or metabolic disturbances;
* Has unstable cardiovascular disease, defined as a recent clinical deterioration (e.g., unstable angina, rapid atrial fibrillation, or transient ischemic attack) in the last 3 months prior to screening or a cardiac hospitalization within the last 3 months prior to screening;
* Currently has a malignancy or has a history of malignancy within 5 years before screening (with the exception of a nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study agent administration or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before the first Guselkumab administration);
* Has a history of lymphoproliferative disease, including lymphoma; a history of monoclonal gammopathy of undetermined significance; or signs and symptoms suggestive of possible lymphoproliferative diseases, such as lymphadenopathy or splenomegaly;
* Has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (e.g., bronchiectasis), recurrent urinary tract infection (e.g., recurrent pyelonephritis or chronic nonremitting cystitis), fungal infection (e.g., mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers;
* Has a transplanted organ (with exception of a corneal transplant >3 months before the first administration of the study agent);
* Has a history of an infected joint prosthesis, or has ever received antibiotics for a suspected infection of a joint prosthesis, if that prosthesis has not been removed or replaced;
* Has or has had a serious infection (e.g., sepsis, pneumonia, or pyelonephritis) or has been hospitalized or received IV antibiotics for an infection within 2 months before screening;
* Has or has had a herpes zoster infection within 2 months before screening;
* Is pregnant, nursing, or planning a pregnancy (both men and women) within 12 weeks after receiving the last administration of the study agent;
* Has received, or is expected to receive, any live virus or bacterial vaccination within 3 months before the first administration of the study agent;
* Has had a BCG vaccination within 12 months of screening;
* Has known intolerance or hypersensitivity to any biologic medication, or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies, or antibody fragments;
* Subject has known allergies, hypersensitivity, or intolerance to Guselkumab or its excipients;
* Has a history of active granulomatous infection, including histoplasmosis or coccidioidomycosis, before screening;
* Has a chest radiograph within 3 months prior to the first administration of the study agent that shows an abnormality suggestive of a malignancy, significant cardiovascular or pulmonary disease, or current active infection, including TB;
* Has ever had a nontuberculous mycobacterial infection or opportunistic infection (e.g., cytomegalovirus, pneumocystosis, aspergillosis);
* Is infected with human immunodeficiency virus (HIV, a confirmed positive serology for HIV antibody);
* Tests positive for hepatitis B virus (HBV) infection at screening; - Is seropositive for antibodies to hepatitis C virus (HCV) at screening, unless the subject had 2 negative HCV ribonucleic acid (RNA) test results at least 6 months apart prior to screening and has a third negative HCV RNA test result at screening;
* Has had major surgery (e.g., requiring general anesthesia and hospitalization) within 8 weeks before the screening, or will not have fully recovered from such surgery, or has such major surgery planned during the time the subject is expected to participate in the study; NOTE: Subjects with planned surgical procedures to be conducted under local anesthesia may participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
pain-related genes mRNA | 6 months
  Change in synovial transcriptomic profiling of pain-related genes (as described by Perkins JR et al, Pain 2013; Bratus-Neuenschwander A et al, Genes 2018) in PsA patients before and after six months of treatments with Guselkumab.

CONTACTS AND LOCATIONS:
Locations (1):
- Immunorheumatology Unit, Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Italy, Italy